CLINICAL TRIAL: NCT00700869
Title: Phase 2 Study of a New Mechanical Ventilation Weaning Strategy Governs by a Respiratory Behaviour Status Assessment for Patients With Altered Level of Consciousness
Brief Title: Evaluation of a New Mechanical Ventilation Weaning Strategy for Patients With Altered Level of Consciousness
Acronym: ORGAR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P070204
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-09

CONDITIONS: Artificial Respiration; Consciousness Disorders; Wearing Off Effect
Keywords: Altered level of consciousness; Tracheal tube withdrawal; Respiration; Artificial Respiration; Physiology
MeSH Terms: conditions — Consciousness Disorders; Respiratory Aspiration | interventions — Respiration, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Tracheal tube withdrawal governs by respiratory behaviour status
  Interventions: Procedure: mechanical ventilation

INTERVENTIONS:
Procedure: mechanical ventilation — mechanical ventilation

SUMMARY:
The purpose of this study is to determine if a weaning strategy from artificial ventilation governs by respiratory behaviour status assessed by our method is safe enough.

DETAILED DESCRIPTION:
Current guidelines for mechanical ventilation weaning do not apply for patients with altered level of consciousness. One major limitation is a failure of clinical assessment of the respiratory behaviour status of these patients that are not able to interact appropriately with the examiner. We propose a non-invasive method for the respiratory behaviour assessment of a patient under artificial ventilation that do not requires his participation. Our hypothesis is that, in case of normal respiratory behaviour status, it is possible to wean under security a patient despite his abnormal level of consciousness.We previously demonstrate that patients successfully wean by the clinical team also disclose a normal respiratory behaviour status while patients with weaning failure had abnormal respiratory behaviour. In the present study, we wonder to evaluate that a weaning strategy governs by respiratory behaviour status assessed by our method is safe. For this purpose, in this study, tracheal tube withdrawal is triggered by a recognition of a normal respiratory behaviour status assessed daily in patients under mechanical ventilation with an altered level of consciousness and a good tolerance to T tube challenge.

ELIGIBILITY:
Inclusion Criteria:

* Altered level of consciousness (-1 < RASS > +1)
* Mechanical ventilation ( > 72 hours)
* Withdrawal of sedative drugs (> 48 hours)
* T tube challenge tolerance
* Signed approval for the study by close relative or legal representative

Exclusion Criteria:

* Respiratory disease prior to the actual artificial ventilation requirement.
* Impairment of upper airway function prior to the actual artificial ventilation requirement.
* Pregnancy
* Minor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Rate of successful mechanical ventilation weaning at 72 hours | 72 hours

SECONDARY OUTCOMES:
Post tracheal tube withdrawal pneumonia at 72 hours | 72 hours
Rate of auto-extubation during patient's participation to the protocol | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Laurent HEYER, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Anesthesia and CCM; Lariboisière Hospital, Paris, France